CLINICAL TRIAL: NCT03367338
Title: The Effect of Low-Phosphate Diet on Fibroblast Growth Factor-23 Level in Patients Undergoing Hemodialysis
Brief Title: Low-Phosphate Diet and Fibroblast Growth Factor-23 Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wan-Chuan Tsai (Other)
Responsible Party: Sponsor-Investigator, Wan-Chuan Tsai, Attending Physician, Far Eastern Memorial Hospital
Organization: Far Eastern Memorial Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FEMH-IRB-106108-F
Record Dates: First submitted 2017-12-05; First posted 2017-12-08 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis; Hyperphosphatemia; Dietary Intervention; Elevated Fibroblast Growth Factor-23
MeSH Terms: conditions — Hyperphosphatemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Participants in group A consumed a 2-day very low-phosphate diet with PPR of 8 mg/g, followed by a 5-day washout period in which they adhered to usual diets, and then consumed a 2-day low-phosphate diet with PPR of 10 mg/g.
  Interventions: Other: Low-phosphate diet
- Group B (Active Comparator): Compared with group A, the opposite order of low-phosphate diets will be prescribed in group B.
  Interventions: Other: Low-phosphate diet

INTERVENTIONS:
Other: Low-phosphate diet — Very low-phosphate diet, PPR value of 8 mg/g, vs. low-phosphate diet, PPR value of 10 mg/g

SUMMARY:
The aims of the study are to evaluate the effect of low-phosphate diet on FGF23 level and to determine the optimal amount of dietary phosphate restriction in hemodialysis patients. In particular, the investigators will assess the comparing effect of pre-specified low-phosphate diets, very low-phosphate diet, phosphate-to-protein ratio (PPR) value of 8 mg/g, versus low-phosphate diet, PPR value of 10 mg/g, on the change of FGF23 and phosphate level.

DETAILED DESCRIPTION:
In patients with hemodialysis, the prevalence of cardiovascular disease (CVD) is high, and is the leading cause of death. Among several cardiovascular risk factors of hemodialysis patients, elevated fibroblast growth factor-23 (FGF23) level is common, and plays major role in the development of CVD with independent pathophysiologic mechanisms. Evidence from animal studies demonstrated that low-phosphate diet reduced FGF23 level. Clinical trials assessing the effect of dietary phosphate restriction on FGF23 focused on non-dialysis populution. However, little is known about the effect of low-phosphate diet on FGF23 in hemodialysis patients who have higher prevalence of hyperphosphatemia and severely elevated FGF23 level. In addition, current clinical guideline, based on evidence from observational studies of non-dialysis population, has recommended that dietary phosphate intake should be restricted to 800-1000 mg/day (adjusted for dietary protein needs) when serum phosphate levels are greater than 5.5 mg/dL in those with kidney failure. For hemodialysis population, the optimal amount of dietary phosphate restriction has not been determined. The aims of the study are to evaluate the effect of low-phosphate diet on FGF23 level and to determine the optimal amount of dietary phosphate restriction in hemodialysis patients. In particular, the investigators will compare the effect of pre-specified low-phosphate diets, very low-phosphate diet, phosphate-to-protein ratio (PPR) value of 8 mg/g, versus low-phosphate diet, PPR value of 10 mg/g, on the change of FGF23 and phosphate level.

It is to conduct a randomized, active-controlled trial with cross-over design at a hemodialysis unit of tertiary teaching hospital in Northern Taiwan. Subjects with aged older than 20 years, end-stage renal disease undergoing thrice-weekly hemodialysis for more than three months, having adequate dialysis (urea reduction ratio equal to or greater than 65%) and the most recent serum phosphate level greater than 5.5 mg/dL or between 3.5 and 5.5 mg/dL with regular phosphate binder use will be randomly assigned into two groups: those in group A will receive 2-day diet with known PPR of 8 mg/g, followed by 5-day washout period and then receive another 2-day diet with PPR of 10 mg/g. The opposite order of diets will be prescribed in group B. The study diets will be prepared and cooked at hospital cafeteria. Dietary compositions of the study diets were analyzed before the start of the study. Primary outcome measures are difference in change-from-baseline intact FGF-23 level between the two dietary interventions. Secondary outcomes include changes in serum phosphate, intact parathyroid hormone and C-terminal FGF-23 level.

Since food additives include readily absorbable inorganic phosphorus, only natural food sources were chosen for study diets. All study food items had the following unique characteristics including: 1. Using locally produced raw materials. 2. Meeting healthy and safety requirements. 3. Complying with national quality standards. Prior to enrollment of the eligible patients, the study diets were prepared and cooked with the food hygiene practice using Hazard Analysis and Critical Control Points (HACCP) system at hospital cafeteria and dietary composition of study diets were analyzed for chemical analysis. With reference to Association of Official Analytical Communities (AOAC) Official Method 984.27, phosphorus, and calcium were determined by inductively coupled plasma-optical emission spectrometer (ICP-OES) analysis with the detection limit of 0.1 mg/L. In brief, the sample weight were obtained, the edible portions of samples were ashed at high temperature, digested in nitric acid, and used inductively coupled plasma to determine their actual contents of phosphorus and calcium. With reference to Taiwanese official methods, study diets were measured for analyses of protein, fat, saturated fat, sugar, moisture, and ash. Carbohydrates were calculated by the formula: 100 - (Protein + Fat + Moisture + Ash) (g/100 g). Calories were calculated by the formula: Protein (g) x 4 kcal + Fat (g) x 9 kcal + Carbohydrate (g) x 4 kcal.

Based on the measured values of food items, dietitian had crafted low-phosphate diets. Less than 800 mg per day of phosphate amount is designed to fulfill the current clinical recommendation. Two different contents of phosphate diets were prepared to find out the optimal amount of dietary phosphate. Each of the diets was designed to have similar calcium, protein and total caloric contents but only differ in phosphate contents. To enhance nutrition, and to reduce phosphate amount and bioavailability, study diets were designed to fulfill the following criteria including high protein diet (≧1.2 g/kg/day), adequate calories (≧ 30 kcal/kg/day), low phosphate-to-protein ratio (< 10 mg/g), and higher percentage of plant source of phosphate than that of animal source. In addition, meats were sliced and boiled for 30 minutes before cooking to reduce the amount of phosphate while preserving protein content.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with end-stage kidney disease undergoing thrice-weekly hemodialysis for more than three months, the most recent serum phosphate level greater than 5.5 mg/dL or between 3.5 and 5.5 mg/dL with regular phosphate binder use, and having adequate dialysis (urea reduction ratio equal to or greater than 65%)

Exclusion Criteria:

* Subjects with serum albumin less than 2.5 g/dL, having psychiatric disorders, mental retardation or poor adherence

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-08 (Actual)

PRIMARY OUTCOMES:
Difference in change-from-baseline intact FGF-23 | 2 days
  Difference in change-from-baseline intact FGF-23 level between two low-phosphate diets, very low-phosphate diet, PPR value of 8 mg/g, with low-phosphate diet, PPR value of 10 mg/g

SECONDARY OUTCOMES:
Difference in change-from-baseline serum phosphate | 2 days
  Difference in change-from-baseline serum phosphate level between two low-phosphate diets, very low-phosphate diet, PPR value of 8 mg/g, with low-phosphate diet, PPR value of 10 mg/g
Difference in change-from-baseline intact parathyroid hormone | 2 days
  Difference in change-from-baseline intact parathyroid hormone level between two low-phosphate diets, very low-phosphate diet, PPR value of 8 mg/g, with low-phosphate diet, PPR value of 10 mg/g
Difference in change-from-baseline C-terminal FGF23 | 2 days
  Difference in change-from-baseline C-terminal FGF23 level between two low-phosphate diets, very low-phosphate diet, PPR value of 8 mg/g, with low-phosphate diet, PPR value of 10 mg/g

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Chuan Tsai, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

REFERENCES:
- [Background] Grabner A, Amaral AP, Schramm K, Singh S, Sloan A, Yanucil C, Li J, Shehadeh LA, Hare JM, David V, Martin A, Fornoni A, Di Marco GS, Kentrup D, Reuter S, Mayer AB, Pavenstadt H, Stypmann J, Kuhn C, Hille S, Frey N, Leifheit-Nestler M, Richter B, Haffner D, Abraham R, Bange J, Sperl B, Ullrich A, Brand M, Wolf M, Faul C. Activation of Cardiac Fibroblast Growth Factor Receptor 4 Causes Left Ventricular Hypertrophy. Cell Metab. 2015 Dec 1;22(6):1020-32. doi: 10.1016/j.cmet.2015.09.002. Epub 2015 Oct 1. PMID 26437603
- [Background] Isakova T, Gutierrez OM, Smith K, Epstein M, Keating LK, Juppner H, Wolf M. Pilot study of dietary phosphorus restriction and phosphorus binders to target fibroblast growth factor 23 in patients with chronic kidney disease. Nephrol Dial Transplant. 2011 Feb;26(2):584-91. doi: 10.1093/ndt/gfq419. Epub 2010 Jul 14. PMID 20631407
- [Background] Di Iorio B, Di Micco L, Torraca S, Sirico ML, Russo L, Pota A, Mirenghi F, Russo D. Acute effects of very-low-protein diet on FGF23 levels: a randomized study. Clin J Am Soc Nephrol. 2012 Apr;7(4):581-7. doi: 10.2215/CJN.07640711. Epub 2012 Feb 23. PMID 22362063
- [Background] Tsai WC, Wu HY, Peng YS, Hsu SP, Chiu YL, Chen HY, Yang JY, Ko MJ, Pai MF, Tu YK, Hung KY, Chien KL. Effects of lower versus higher phosphate diets on fibroblast growth factor-23 levels in patients with chronic kidney disease: a systematic review and meta-analysis. Nephrol Dial Transplant. 2018 Nov 1;33(11):1977-1983. doi: 10.1093/ndt/gfy005. PMID 29420827